CLINICAL TRIAL: NCT00611793
Title: A Phase I Trial of PTK787/ZK222584 in Combination With Bevacizumab (Avastin) in Patients With Refractory and/or Advanced Malignancies
Brief Title: PTK787/ZK222584 With Bevacizumab in Patients With Refractory and/or Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Howard A. Burris, III, M.D., SCRI Oncology Research Consortium
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI REFMAL 56
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Refractory Malignancy; Advanced Malignancies
Keywords: Refractory Malignancy; Advanced Malignancies; PTK787/ZK222584; Bevacizumab
MeSH Terms: conditions — Neoplasms | interventions — vatalanib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): PTK787/ZK222584 and Bevacizumab
  Interventions: Drug: PTK787/ZK222584 and Bevacizumab

INTERVENTIONS:
Drug: PTK787/ZK222584 and Bevacizumab — PTK787/ZK222584 will be administered as a single agent orally on days 1-14 of cycle 1. The day 14 dose of PTK787/ZK222584 will be administered in the outpatient clinic and PK samples will be obtained. On Day 15 the patient will receive the initial dose of IV bevacizumab and PTK787/ZK222584. Bevacizumab will be repeated at 2 week intervals in patients with stable disease or better for four cycles of treatment (16 weeks). After four treatment cycles, only patients with a PR or CR will continue treatment with PTK787/ZK222584 and bevacizumab. Patients with stable disease may continue single agent PTK787/ZK22258 from cycle 5 onward. Protocol treatment will continue until disease progression or intolerable toxicity warrants drug discontinuation.

SUMMARY:
PTK787/ZK222584 is an orally active inhibitor of VEGF-R tyrosine kinases. Bevacizumab is an intravenous humanized monoclonal antibody directed against vascular endothelial growth factor. By binding to VEGF, bevacizumab blocks VEGF-A receptor binding. Due to the different mechanisms of action and the non-overlapping toxicity profiles of the two agents, it is hoped that a combination regimen incorporating both compounds will produce increased activity without enhanced toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven advanced solid tumors that are resistant to standard treatment and/or for which there is no known effective therapy
* Age ≥ 18 years old
* ECOG Performance Status of 0 or 1
* Laboratory values ≤ 7 days prior to treatment:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L (≥ 1500/mm3)
  * Platelets (PLT) ≥ 100 x 109/L (≥ 100,000/mm3)
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Serum creatinine ≤ 1.5 ULN
  * Serum bilirubin ≤ 1.5 ULN
  * International Normalized Ratio (INR) <2.0
  * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 3.0 x ULN
  * Negative for proteinuria based on dip stick reading OR, if documentation of +1 result for protein on dip stick reading, then total urinary protein ≤ 500 mg and measured creatinine clearance (CrCl) ≥ 50 mL/min from a 24-hour urine collection
* Life expectancy ≥ 12 weeks
* Written informed consent obtained according to local guidelines

Exclusion Criteria:

* History or presence of central nervous system (CNS) disease (i.e., primary brain tumor, malignant seizures, CNS metastases or carcinomatous meningitis)
* Patients with a history of another primary malignancy ≤ 5 years, with the exception of inactive basal or squamous cell carcinoma of the skin
* Prior chemotherapy ≤ 3 weeks prior to registration and/or randomization. Patients must have recovered from all therapy-related toxicities
* Prior biologic or immunotherapy ≤ 2 weeks prior to registration and/or randomization. Patients must have recovered from all therapy-related toxicities
* Prior full field radiotherapy ≤ 4 weeks or limited field radiotherapy ≤ 2 weeks prior to randomization. Patients must have recovered from all therapy-related toxicities. The site of previous radiotherapy should have evidence of progressive disease if this is the only site of disease
* Major surgery (i.e., laparotomy) ≤ 4 weeks prior to randomization. Minor surgery ≤ 2 weeks prior to randomization. Insertion of a vascular access device is not considered major or minor surgery in this regard. Patients must have recovered from all surgery-related toxicities
* Patients who have received investigational drugs ≤ 4 weeks prior to registration and/or randomization
* Prior therapy with anti-VEGF agents (including PTK787/ZK222584 and bevacizumab)
* Pleural effusion or ascites that causes respiratory compromise (≥ CTC grade 2 dyspnea)
* Female patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control. Barrier contraceptives must be used throughout the trial in both sexes. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Women of childbearing potential must have a negative serum pregnancy test 48 hours prior to administration of study treatment. Please refer to appendix 3 for a list of examples of substrates of human liver microsomal P450 enzymes
* Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:

  * Uncontrolled high blood pressure (>160/100 on medication), history of labile hypertension, or history of poor compliance with an antihypertensive regimen
  * Unstable angina pectoris
  * Symptomatic congestive heart failure
  * Myocardial infarction ≤ 6 months prior to registration
  * Serious uncontrolled cardiac arrhythmia
  * Uncontrolled diabetes
  * Active or uncontrolled infection
  * Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* Chronic renal disease
* Acute or chronic liver disease (e.g., hepatitis, cirrhosis)
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PTK787/ZK 222584 (i.e., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow the tablets)
* Patients with confirmed diagnosis of human immunodeficiency virus (HIV) infection are excluded at the investigator's discretion if he/she feels that 1) a potential drug interaction between PTK787/ZK 222584 and any of the patient's anti-HIV medications could influence the efficacy of the anti-HIV medication, or 2) it may place the patient at risk due to the pharmacologic activity of PTK787/ZK 222584. Please refer to appendix 3 for a list of examples of substrates of human liver microsomal P450 enzymes
* Patients who are taking therapeutic warfarin sodium (Coumadin) or similar oral anticoagulants that are metabolized by the cytochrome P450 system. Heparin is allowed. Please refer to appendix 3 for a list of examples of substrates of human liver microsomal P450 enzymes
* Patients receiving chronic daily treatment with aspirin (> 325 mg/day) or with daily doses of platelet inhibitory non-steroidal anti-inflammatory agents (e.g. Ibuprofen 800 mg qid, naproxen 500 mg bid)
* Patients receiving chronic steroid therapy
* Any nonhealing wound, ulcer, or long bone fracture
* Clinical history of hemoptysis or hematemesis within the past 3 months
* Clinical evidence or history of a bleeding diathesis or coagulopathy
* History of stroke within 6 months
* Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-10; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Burris, III, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States